CLINICAL TRIAL: NCT04275986
Title: A Phase II Clinical Trial of Concurrent Chemoradiotherapy After Endoscopic Resection for Stage I Esophageal Squamous Cell Carcinoma
Brief Title: Concurrent Chemoradiotherapy After Endoscopic Resection for Stage I Esophageal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zhouguang Hui, M.D., Chief physician, Director of VIP Department, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19/313-2097
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal Squamous Cell Carcinoma; Endoscopic resection; Concurrent chemoradiotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Radiotherapy, Intensity-Modulated; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Enrolled Patients will receive concurrent chemoradiotherapy per protocol. The radiotherapy clinical target volume will include 2 cm above and below the tumor bed and high-risk lymph nodal area. Intensity modulated radiotherapy techniques will be used with a total dose of 45Gy in 25 fractions. Chemotherapy will be conducted weekly up to 5 weeks. The specific chemotherapy regimen are Paclitaxel Liposome 45mg/m2, d1 and Nedaplatin 25mg/m2, d1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Endoscopic resection+ concurrent chemoradiotherapy
  Interventions: Procedure: Intensity modulated radiotherapy (IMRT); Drug: Chemotherapy

INTERVENTIONS:
Procedure: Intensity modulated radiotherapy (IMRT) — Intensity-modulated radiation therapy (IMRT) with a total dose of 45Gy in 25 fractions
Drug: Chemotherapy — Nedaplatin 25 mg/m2 and Paclitaxel liposome 45mg/m2, day 1, every week, 5 weeks

SUMMARY:
This is a prospective single-arm study of endoscopic resection (ER) following concurrent chemoradiotherapy for stage I esophageal squamous cell carcinoma, to find if the treatment combination is useful by assessing its safety and efficacy.

DETAILED DESCRIPTION:
The objectives are to evaluate the efficacy and safety of concurrent chemoradiotherapy after endoscopic resection in early stage esophageal squamous cell carcinoma by evaluating the effectiveness, including 3-year OS, DFS, LRFS, DMFS, LCR, DMR and QOF, and analyzing the toxicity and side effects in 3 years follow-up time.

The study preliminarily explored the recurrence patterns of solely ER for early esophageal squamous cell carcinoma with high risk factors, analyzed the rationality of target areas and dose choices in the treatment regimen of concurrent chemoradiotherapy after ER, and proposed modification schemes of the target area and dose of radiotherapy. Prospectively acquired hematological samples and tissue samples during the treatment will be tested for genetic testing, single-cell genome sequencing, transcriptome and epigenomic analysis, to screen the population with high risk of recurrence or the population who will benefit from this treatment combination.

In terms of sample size, The estimates of survival rate at 3 years for operation group is 85.1% (95% CI: 82.0%, 87.7%) based on SEER study. Assuming that the survival rate at 3 years for ER+CRT is about 90.7%. The difference between operation and ER+CRT is marginal and clinically meaningless. In our study, we will target to establish that the ER+CRT is non-inferiority to operation in term of survival rate at 3 years, and further investigate the benefit of ER+CRT in safety profile and quality of life. A non-inferiority margin 10% is applied with respect to 85.1%. A number of 50 subjects is adequate to achieve 80% statistical power under a type one error rate 0.025 one-sided. The power analysis is based on simulation, 10000 iterations are carried out, Greenwood's method is applied.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 to 75 years (18 years and 75 years are inclusive).
* The Eastern Cooperative Oncology Group (ECOG) performance status score is 0 to 1 point.
* Weight loss (intentional or unintentional) of less than or equal to 10% of body weight in the 6 months prior to surgery.
* Complete radiological staging is required before ER, including gastroscopy, endoscopic ultrasonography, chest CT, brain MRI and bone scan (if positive, bone metastasis must be confirmed by MRI or CT examination of corresponding parts, otherwise bone metastasis cannot be determined). No lymph nodes with shorter diameter >10mm in mediastinum presented by endoscopic ultrasonography or chest CT. No abdominal nor neck lymph node metastases presented by B-ultrasound.
* Primary lesion located in thoracic esophagus.
* Clinical stage: cT1（sm1/sm2）N0M0 (The 8th edition of American Joint Committee on Cancer [AJCC]) before ER.
* ER is a complete removal of tumor.
* Pathologically confirmed squamous cell carcinoma.
* Histologically confirmed diagnosis of T1a with LVI, T1b（sm1/sm2）with/without LVI, or microscopically positive vertical resection margin (R1 resection).
* Less than three endoscopically resected synchronous lesions with high risk factors (lymphovascular or mucous membrane invasion, submucous infiltration, poor differentiation or microscopically positive vertical resection margin), which can be safely encompassed in a tolerable radiation plan.
* Non-pregnancy and non-pregnancy plan in the next 12 months (urine pregnancy test or blood pregnancy test is required for women of childbearing age to exclude pregnancy).
* No serious medical disease nor organ dysfunction. Adequate BM, liver, kidney and heart function.
* Meet the treatment and follow-up criteria, able to receive treatment, follow-up and pathological examination. The subject has voluntarily signed the written informed consent form (ICF).

Exclusion Criteria:

* Any positive N or M stage.
* Macroscopic residual tumor (R2 resection).
* Lesions with poor prognistic factors (lymphovascular or mucous membrane invasion, submucous infiltration, poor differentiation or microscopically positive vertical resection margin) solely resected endoscopically more than six months before evaluation.
* Patients with other malignant tumors within 5 years before enrollment.
* Unavailable gastroscope due to esophageal stenosis.
* Previously received electrocoagulation, other treatments (including photodynamic therapy, multipolar electrocoagulation, argon plasma coagulation, laser therapy, et al.) or radiotherapy.
* Previously received any esophageal surgery, excluding fundoplication with no complications (no slippage, dysphagia, et al.).
* Uncontrolled coagulation disorders: INR >2 or PLT<75,000/μL.
* Patients who are taking or have taken (within 7 days before/after treatment) aspirin, clopidogrel or other non-steroidal anti-inflammatory drugs.
* Patients with history of uncontrolled drug or alcohol dependence that limits the ability to understand or comply with medical orders, including inability to understand and execute ICF, post-treatment orders, or follow-up guidelines.
* Patients implanted pacemakers, including AICD, nerve stimulator or cardiac pacemaker, without the permission from specialist in charge.
* Patients with mental disease, serious medical disease or major organ dysfunction.
* Pregnant, lactating women or women without offspring.
* Patients unable to understand/express informed or consent.
* Patients with known allergy to platinum compounds or paclitaxel.
* Other circumstances which are considered by the investigator that the subject is unsuitable to be enrolled

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 3-year
  OS was defined as the time from endoscopic resection to the last follow-up time or death due to any cause.
Adverse events (AE) | 3-year
  An AE was defined as any untoward medical occurrence in a participant administered study treatment and which did not necessarily have to have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Disease Free Survival (DFS) | 3-year
  DFS was defined as the time from the date of endoscopic resection to the date of tumor recurrence as assessed by RECIST 1.1, the last follow-up or death.
Local Recurrence Free Survival (LRFS) | 3-year
  LRFS was defined as the time from the date of endoscopic resection to the date of local recurrence (Local recurrence: documented evidence of newly found lesions at the primary surgical site and 1 cm around) as assessed by RECIST 1.1, the last follow-up or death.
Disease Metastasis Free Survival (DMFS) | 3-year
  DMFS was defined as the time from the date of endoscopic resection to the date of tumor metastasis as assessed by RECIST 1.1, the last follow-up or death.
Local Control Rate (LCR) | 3-year
  LCR was defined as percentage of participants who did not have local recurrence as assessed by RECIST 1.1 from the date of endoscopic resection to the date of the last follow-up or death.
Distant Metastasis Rate (DMR) | 3-year
  DMR was defined as percentage of participants who had tumor distant metastasis as assessed by RECIST 1.1 from the date of endoscopic resection to the date of the last follow-up or death.
Quality of Life (QOL): questionnaires | 3-year
  Evaluate the quality of life via questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No